CLINICAL TRIAL: NCT05974072
Title: A Feasibility Study of a Multidisciplinary Treatment for Patients with Chronic Low Back Pain: PAINDOC Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Marc Terradas Monllor, Principal Investigator, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAINDOC
Record Dates: First submitted 2023-07-11; First posted 2023-08-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Chronic Low-back Pain
Keywords: chronic pain; pain catastrophizing; therapeutic patient education; therapeutic exercise; mindfulness; cognitive behavioural therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two armed, parallel groups, single blind, unicentric, randomized feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Pharmacological Control) (Active Comparator): The subjects in the control group will be treated following a pharmacological approach according to the latest clinical guidelines for patients with chronic low back pain. Thus, the pharmacological options to be considered in each patient will be those included in the first and second analgesic steps of the WHO (preferably without including minor opioids).
  Interventions: Drug: Usual Care
- PAINDOC Program (Experimental): The PAINDOC Program is a multidisciplinary treatment that integrates four parts provided by different health professionals and consists of 8 sessions carried out in the pain unit of the Hospital Clinic of Barcelona over two months.
  It consists of a therapeutic education (Empowered Relief) session given by a physician from the unit, a pain psychology session given by a psychologist, an introductory mindfulness meditation session given by an advanced practice nurse, and two pain neuroscience education sessions and three therapeutic exercise sessions given by a physiotherapist. This program is already part of the pain unit's routine care practice, so it is considered that the sessions of this program do not represent an additional and specific visit for the patients.
  Interventions: Other: PAINDOC Program

INTERVENTIONS:
Drug: Usual Care — The pharmacological treatment will be individualised according to pain intensity, contraindications and the appearance of adverse effects.
  Other Names: Pharmacological Control
  Arms: Usual Care (Pharmacological Control)
Other: PAINDOC Program — The PAINDOC Program consists in:
  * Therapeutic education: The therapeutic education block consists of two parts: an education session called Empowered Relief (ER) and two pain neuroscience education (NDT) sessions.
  * Psychotherapy: The psychotherapy part consists of one group session of one hour, face-to-face and with groups of up to 15 people, given by the psychologist of the pain unit.
  * Mindfulness Meditation: The Mindfulness Meditation consists of one group session of one hour, face-to-face and with groups of up to 15 people. These are given by a nurse from the pain unit. T
  * Therapeutic exercise: The therapeutic exercise module consists of three sessions of one hour each, face-to-face, with small groups of between 6 and 10 patients, and given by the physiotherapist of the pain unit.
  Other Names: Multidisciplinary and multimodal intervention
  Arms: PAINDOC Program

SUMMARY:
The present feasibility study aims to evaluate the feasibility and adequacy of a multidisciplinary treatment program as a therapeutic option for patients with chronic low back pain referred to the pain unit of the Hospital Clinic of Barcelona. Secondarily, the present study will also evaluate the effect on pain-related outcomes to estimate the number of needed participants for a full trial.

The main questions it aims to answer are:

* Is the proposed multidisciplinary treatment feasible and adequate for chronic low back pain patients?
* Is the proposed multidisciplinary treatment effective in improving pain-related outcomes?

Participants will receive either usual care (pharmacological control) or eight multidisciplinary sessions within two months, composed of therapeutic patient education, mindfulness relaxation, cognitive-behavioural therapy and therapeutic exercise. Besides, participants will be assessed using written questionnaires before and after treatment and two months after treatment.

Researchers will assess the feasibility of the multidisciplinary treatment group and will compare both groups to see if there is any difference in several pain-related outcomes.

DETAILED DESCRIPTION:
Despite improving pharmacological and surgical medical treatment options, long-lasting low back pain is the most frequent pain disorder and a leading cause of disability. Over the past decades, clinicians have acknowledged that a broader view of disease and disability is needed in chronic conditions treatment. Therefore, biological, psychological and social factors must be addressed to improve such conditions.

The present study aims to evaluate the viability and adequacy of a multidisciplinary treatment program (PAINDOC Program) as a therapeutic option for patients with chronic low back pain referred to the pain unit of the Hospital Clínic of Barcelona. The secondary objectives are to evaluate the effect of the PAINDOC Program on the reduction of pain intensity, the improvement of pain-related disability, the improvement of quality of life, and the reduction of pain catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary chronic low back pain (non-specific chronic low back pain).
* Predominantly axial pain, for at least 50% of the time during the last 6 months.
* Average pain intensity equal or greater than 4 out of 10 on a verbal numerical scale, during the present week.
* Predisposed to receive an active, non-pharmacological and non-surgical treatment.

Exclusion Criteria:

* Inflammatory low back pain.
* History of cancer in the past 5 years.
* Unexplained and involuntary weight loss of 10 Kg during the last year.
* Problems in the control of bowel and bladder function.
* Difficulty attending sessions due to severe physical disability.
* Diagnosis of severe mental illness (schizophrenia, major depression, bipolar disorder, etc.).
* Addiction disorder to parenteral drugs or strong prescription opioids. Technical-logistical problems (inability to attend treatment sessions, inability to complete evaluation questionnaires).
* Seeking compensation or litigation in the last year.
* Severe hearing loss or severe cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 4 months prior to study start
  To obtain this information, the number of participants included in the program for four consecutive months will be calculated. The number of eligible participants, the number of participants included and excluded, and the reasons for exclusion will be detailed.
Number of participants completing treatment | 2 months
  Acceptable compliance has been defined as at least 80% of participants included in the program completing all program sessions.
Follow-up rate | 4 months
  to determine the follow-up rate, the number of participants who complete the evaluations at each evaluation point in the study will be detailed.
Acceptance of treatment and detection of barriers | 2 months
  Treatment acceptance will be assessed through a qualitative approach, based on focus groups and content analysis. The study will have a phenomenological approach to understand and know directly the experiences of the participants. The research will be conducted from the interpretive paradigm, as it seeks to understand and interpret the deep meaning of the observed phenomena. In addition, it is based on an inductive methodology that starts from reality to generate theories, so the fieldwork does not start from a hypothesis.

SECONDARY OUTCOMES:
Pain Intensity. Changes from baseline to 2 months after treatment. | Baseline, 2 months, 4 months
  Participants will be asked to rate their pain intensity on a horizontal 100-mm Visual Analogue Scale (VAS), ranging from 0 = no pain to 100 = worst imaginable pain. The VAS is a valid and reliable instrument compared with other pain rating scales, and has been well established in clinical practice and research for measuring pain levels in low back pain patients. For patients with subacute or chronic low back pain, the minimum clinically relevant change is considered to be at least 20 mm on a VAS.
Pain-related disability. Changes from baseline to 2 months after treatment. | Baseline, 2 months, 4 months
  Disability will be assessed using the spanish version of the Oswestry Disability Index (ODI) questionnaire. The ODI is one of the most common specific measurement tools to evaluate the function and disability of lumbar spine pathologies. This questionnaire contains 10 items evaluated from 0 to 5 (higher values indicate greater disability), which correspond to 10 domains. The sum of the 10 scores is expressed as a percentage (ODI score), with ranges from 0% (no disability) to 100% (maximum disability).
Health-related quality of life. Changes from baseline to 2 months after treatment. | Baseline, 2 months, 4 months
  The spanish version of the Euro Quality of Life 5D-5L (EQ-5D-5L) was used to assess the health related quality of life (HRQL).(10) The EQ-5D-5L consists in two pages: the first one is based on a descriptive system that defines health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories: no problems, slight problems, moderate problems, severe problems, extreme problems.(10) A health state is composed by taking one level for each dimension, and a preference-based scoring function is used to convert the descriptive system to a summary index score (ranging from states worse than dead <0 to full health 1).
Pain Catastrophizing. Changes from baseline to 2 months after treatment. | Baseline, 2 months, 4 months
  The Spanish version of Pain Catastrophizing Scale (PCS) was used to asses thoughts and feelings related to pain experiences.(9) The PCS is a 13 item self-administered questionnaire composed of 3 subscales: rumination, magnification and helplessness. The PCS uses a 5-point Likert scale with responses ranging from 0 = not at all to 4 = all the time. Overall scores range from 0 to 52 points, the higher the score, the higher is the pain catastrophism level.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143
- [Background] Darnall BD, Roy A, Chen AL, Ziadni MS, Keane RT, You DS, Slater K, Poupore-King H, Mackey I, Kao MC, Cook KF, Lorig K, Zhang D, Hong J, Tian L, Mackey SC. Comparison of a Single-Session Pain Management Skills Intervention With a Single-Session Health Education Intervention and 8 Sessions of Cognitive Behavioral Therapy in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2113401. doi: 10.1001/jamanetworkopen.2021.13401. Erratum In: JAMA Netw Open. 2022 Apr 1;5(4):e229739. doi: 10.1001/jamanetworkopen.2022.9739. PMID 34398206
- [Derived] Dalmau-Roig A, Dursteler C, Ochandorena-Acha M, Vilchez-Oya F, Martin-Villalba I, Obach A, Terradas-Monllor M. A multidisciplinary pain management program for patients with chronic low back pain: a randomized, single-blind, controlled, feasibility study. BMC Musculoskelet Disord. 2025 Jan 17;26(1):59. doi: 10.1186/s12891-025-08294-8. PMID 39825315